CLINICAL TRIAL: NCT04979429
Title: Preventing Chronic Post-Surgical Pain and Prolonged Opioid Use: The Perioperative Pain Self-Management Program
Brief Title: The Perioperative Pain Self-Management Program Trial
Acronym: PePS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IIR 20-115
Record Dates: First submitted 2021-07-15; First posted 2021-07-28 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; opioid
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either receive the pain self-management sessions (PePS) or standard care (SC).
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to randomization status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PePS (Experimental): 4 sessions of telephone CBT-based pain self-management in addition to standard perioperative care.
  Interventions: Behavioral: Perioperative Pain Self-management (PePS)
- Standard Care (No Intervention): Standard perioperative care.

INTERVENTIONS:
Behavioral: Perioperative Pain Self-management (PePS) — 4 sessions of telephone CBT-based pain self-management.
  Other Names: PePS
  Arms: PePS

SUMMARY:
This study will trial the impact of teaching surgical patients a pain self-management approach to compliment medical post-surgical pain management.

DETAILED DESCRIPTION:
Surgery can precipitate the development of both chronic pain and long-term opioid use. There is a need for strategies to augment perioperative pharmacotherapeutic management of pain with non-pharmacologic strategies to prevent long-term sequelae. Psychological interventions such as cognitive behavioral therapy (CBT) can effectively reduce distress and improve functioning among patients with chronic pain. While CBT has been used extensively in patients with established chronic pain, it has not been used as a preventive intervention targeting the transition from acute to chronic postsurgical pain. The Perioperative Pain Self-management (PePS) program has the potential to reduce the incidence of chronic post-surgical pain and long-term opioid use among Veterans. This study will: Examine the efficacy of PePS compared to standard care on 6-month pain (primary outcome), mood and functioning outcomes as well as time to post-surgical opioid and other analgesic use cessation.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for total hip, knee, or shoulder joint arthroplasty through the Iowa City, IA, Des Moines, IA, Minneapolis, IA, or Milwaukee WI, VA medical centers

Exclusion Criteria:

* inability to complete study forms/procedures because of a language/literacy barrier
* active bipolar or psychotic disorder
* history of brain injury
* dementia
* CBT therapy within the past year
* lack of access to a telephone for PePS sessions

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 6-months post-surgery
  Surgical Site Pain
  The Numeric Rating Scale (NRS) is a 0-10 measure where 0 = no pain.

SECONDARY OUTCOMES:
opioid use | time to cessation post surgery (weekly phone calls for the first 6 weeks)
  Time to opioid cessation following surgery: daily opioid use will be collected via weekly phone calls for the first 6 weeks post-surgery.

OTHER OUTCOMES:
Patient Health Questionnaire 8-item version (PHQ-8) | Change between pre-surgery and 6-months post-surgery
  A measure of depressive symptoms. Scores range from 0-24 with higher scores indicating more depressive symptoms.
General Anxiety Disorder Scale: 7-item (GAD-7) | Change between pre-surgery and 6-months post-surgery
  A measure of anxious symptoms. Scores range from 0-21 with higher scores indicating more anxious symptoms.
Pain Disability Index (PDI) | Change between pre-surgery and 6-months post-surgery
  A measure of pain-related functioning. Scores range from 0-70 with higher scores indicating greater pain-related disability.
Brief pain inventory | 6 months post-surgery
  Generalized body pain intensity and pain interference. Scores range from 0-10 with higher scores indicating more pain severity and interference.
Other analgesic use | time to cessation post-surgery (weekly phone calls for the first 6 weeks post-surgery)
  Time to cessation of other analgesics following surgery: daily analgesic use will be collected via weekly phone calls for the first 6 weeks post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine E Hadlandsmyth, PhD MA MS, Principal Investigator — Iowa City VA Health Care System, Iowa City, IA
Locations (2):
- United States (2):
  - Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hadlandsmyth K, Burgess DJ, Leparski RF, Odom AS, Campbell EJ, Obrecht AA, Adamowicz JL, Cho H, Steffensmeier KS, Johnson NL, Richards CC, Vander Weg MW, Lund BC, Yoon P, Mosher HJ. The Perioperative Pain Self-Management (PePS) randomized controlled trial protocol: Preventing chronic post-surgical pain and prolonged opioid use. Contemp Clin Trials. 2022 Jul;118:106810. doi: 10.1016/j.cct.2022.106810. Epub 2022 May 31. PMID 35660486

DOCUMENTS (1):
  • Informed Consent Form (2023-12-21): https://cdn.clinicaltrials.gov/large-docs/29/NCT04979429/ICF_000.pdf